CLINICAL TRIAL: NCT05307913
Title: EIT-guided PEEP Titration Versus Low PEEP/FiO2 Table for ARDS: a Multicenter, Randomized, Controlled Trial
Brief Title: PET - PEEP by EIT for Acute Respiratory Distress Syndrome Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEEP by EIT for ARDS
Record Dates: First submitted 2021-12-29; First posted 2022-04-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2022-04

CONDITIONS: ARDS, Human
Keywords: electrical impedance tomography; ARDS; PEEP
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT-guided PEEP (Experimental): PEEP titration by EIT
  Interventions: Other: EIT-guided PEEP
- Table-guided PEEP (Active Comparator): PEEP selection by the lower PEEP/FiO2 table
  Interventions: Other: Table-guided PEEP

INTERVENTIONS:
Other: EIT-guided PEEP — PEEP setting according to EIT
  Arms: EIT-guided PEEP
Other: Table-guided PEEP — PEEP setting according to the lower PEEP/FiO2 table
  Arms: Table-guided PEEP

SUMMARY:
This study is a multicentric randomized controlled study.The objective of this study is to compare the prognosis of patients with ARDS between EIT-oriented individualized PEEP and traditional lower PEEP/FiO2 table-oriented PEEP strategy.

ELIGIBILITY:
Inclusion Criteria:

Intubated, mechanically ventilated patients with diagnosis of ARDS according to ARDS Berlin standard by attending doctor

Exclusion Criteria:

1. Age < 18 years old and > 90 years old;
2. Pregnancy;
3. EIT contradictions (presence of pacemaker or automatic implantable cardioverter defibrillator);
4. Severe intracranial hypertension;
5. Pneumothorax, pneumomediastinum, subcutaneous emphysema or at high-risk for pneumothorax (e.g., pneumatocele, interstitial lung disease);
6. Unstable hemodynamic status intorerable to lung recruitment and PEEP titration, judged by an attending intensivist; (This may be a transient criterion, since patients meeting this criterion might be included later if hemodynamics improves)
7. End status of disease;
8. Patients or their families refused to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Survival in 28 days | 28 days
  Survival within 28 days from randomization

SECONDARY OUTCOMES:
Lenght of ICU stay | Maximum 6-months
  Length of hospital stay from randomization to ICU discharge
Lenght of hospital stay | Maximum 6-months
  Length of hospital stay from randomization to hospital discharge
28-day ventilator-free days | 28 days
  Number of days alive and out of mechanical ventilation between randomization and 28 days after randomization.
Barotrauma | 7 days
  We consider as barotrauma within 7 days any pneumothorax, pneumomediastinum, subcutaneous emphysema or pneumatocele > 2cm detected on image exams between randomization and 7 days, except those judged to be clearly caused by invasive procedures.
ICU survival | Maximum 6-months
  Survival at ICU discharge.
hospital survival | Maximum 6-months
  Survival at hospital discharge.
change of Sequential Organ Failure Assessment (SOFA) score | 2 days
  change of SOFA score within first 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong H, Chi Y, Zhang R, Yin C, Jia J, Wang B, Liu Y, Shang Y, Wang R, Long Y, Zhao Z, He H. Multicentre, parallel, open-label, two-arm, randomised controlled trial on the prognosis of electrical impedance tomography-guided versus low PEEP/FiO2 table-guided PEEP setting: a trial protocol. BMJ Open. 2024 Feb 1;14(2):e080828. doi: 10.1136/bmjopen-2023-080828. PMID 38307528